CLINICAL TRIAL: NCT00002238
Title: Phase III Randomized Double-Blind Placebo Controlled Study To Evaluate the Safety and Efficacy of Betaseron in AIDS and Advanced ARC Patients Receiving a Reduced-Dose AZT Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 002A; TBO1-310188
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Interferon Type I
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Interferon beta-1b; Zidovudine

INTERVENTIONS:
Drug: Interferon beta-1b
Drug: Zidovudine

SUMMARY:
To evaluate the safety and efficacy of interferon beta (Betaseron) in AIDS and advanced AIDS related complex (ARC) patients receiving a reduced-dose zidovudine (AZT) regimen.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).

Patient must have:

* Uninterrupted therapy with reduced-dose AZT 500 - 600 mg/day for at least 3 weeks before entry.
* Acceptable hepatic and renal function.
* AMENDED to delete the following sentence:
* Hematologic intolerance to full-dose zidovudine (AZT) (1000 - 1200 mg/day).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Concurrent, ineffectively controlled opportunistic infections.
* Extensive cutaneous and/or visceral Kaposi's sarcoma requiring systemic chemotherapy.
* Proteinuria of 2+ or greater.
* HIV encephalopathy.
* HIV wasting syndrome.
* New York Heart Classification III or IV.
* Uncontrolled angina pectoris.
* Evidence of clinically significant, multifocal uncontrolled cardiac dysrhythmias.

Concurrent Medication:

Excluded:

* Antiretrovirals other than zidovudine (AZT) or Betaseron.
* Chronic acyclovir therapy.
* Acetaminophen.

Patients with the following are excluded:

* Intolerance (hematologic or otherwise) to zidovudine (AZT) at a dose of 100 mg orally every 4 hours. AMENDED to:
* Intolerance at a dose of 500 to 600 mg/day.
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or complete the study.

Prior Medication:

Excluded within 30 days of study entry:

* Cytotoxic chemotherapy.
* Prior therapy with alpha, beta, or gamma interferons.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Alta Bates / Herrick Hosp, Berkeley, California
  - USC School of Medicine / Norris Cancer Hosp, Los Angeles, California
  - Cedars Sinai Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Summitt Med Ctr / San Francisco Gen Hosp, Oakland, California
  - UCI Med Ctr, Orange, California
  - Davies Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Dr William Davis, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of South Florida, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Chelsea Village Med Ctr, New York, New York
  - Dr Douglas Dieterich, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Thomas Jefferson Med College, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Graduate Hosp, Philadelphia, Pennsylvania
  - Univ TX Galveston Med Branch, Galveston, Texas